CLINICAL TRIAL: NCT02112929
Title: Regional Lung Imaging and Modelling to Quantify Anatomy, Ventilation and Perfusion Using Hyperpolarized Xenon Gas MR and Thoracic CT Imaging
Brief Title: Regional Lung Imaging Using Hyperpolarized Xenon Gas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Oxford University Hospitals NHS Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); University of Sheffield (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HPX-2011-001; 2011-002027-17 (EudraCT Number)
Record Dates: First submitted 2012-07-10; First posted 2014-04-14 (Estimated); Last update posted 2022-02-23 (Actual); Status verified 2021-10

CONDITIONS: Lung Disease
Keywords: Magnetic Resonance Imaging; Lung Diseases
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Inhalation of hyperpolarized xenon (Experimental): One litre of hyperpolarized xenon to be inhaled during MRI scan of the lungs
  Interventions: Drug: Hyperpolarized xenon

INTERVENTIONS:
Drug: Hyperpolarized xenon — Inhalation of up to one litre of polarized xenon gas, up to four inhalations per day are permitted.

SUMMARY:
The investigators aim to use hyperpolarized xenon gas magnetic resonance imaging (MRI) and computed tomography to develop a new technique capable of objectively and quantitatively describing regional and structural lung abnormality. Since this is a relatively novel technique, the investigators first need to acquire imaging and clinical data from a group of participants with normal lungs. The investigators hope to generate an "atlas" of normality, which will form the foundation of future studies to compare with patients suffering from chronic respiratory disease. The investigators also aim to validate the new technique in terms of intra-subject reproducibility.

DETAILED DESCRIPTION:
Currently, the gold standard for assessment of lung function in chronic respiratory disease is spirometry. This is combined with anatomical imaging (chest x-ray and computed tomography) for structural assessment. Spirometry only measures global lung function. It provides no information regarding the different regions of the lung or about the supporting "framework" of the lung itself, the parenchyma. In addition, changes in lung function as measured with spirometric indices do not correlate coherently with the symptoms experienced by patients, nor reflect their decline in health. This weak relationship is probably because the lung is a complex regional organ where localized disturbances of a variety of factors including gas flow (ventilation), blood flow (perfusion) and gas transfer all combine to impair respiratory function.

MRI has the advantage of being an imaging technique free from ionizing radiation making it safe and practical for diseases such as asthma and obstructive lung disease where repeated follow-up scans are necessary. Hyperpolarized xenon, in the doses given for imaging has been shown to be safe. Conventional MRI has limited use in respiratory disease, because the lung is largely composed of air spaces that do not generate an MR signal. Hyperpolarized noble gases can resolve this problem.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male, aged > 18 years.
* Patients with previous histologically verified testicular germ cell tumour who have successfully undergone resection and do not and have never had metastatic disease.
* Normal chest CT, confirmed subjectively by a Consultant Thoracic radiologist (Dr F. Gleeson or R. Benamore or their nominated representative), and no evidence of emphysema on CT density mapping to have been performed no more than one year prior to proposed hyperpolarized Xe-129 MR scan.
* Normal spirometry indices (>80% predicted FEV1 [forced expiratory volume in one second]for age and height) and normal arterial oxygen saturations (SaO2), normal carbon monoxide transfer factor, and generally in good health with no subjective exercise limitation.
* Current non-smokers with no significant smoking history (≤10 pack years) and no history of respiratory disease.
* WHO performance status 0.
* Able (in the Investigators opinion) and willing to comply with all study requirements.
* Willing to allow his General Practitioner and consultant, if appropriate, to be notified of participation in the study.

Exclusion Criteria:

* Inability to give written informed consent.
* Patients with a history of nodal or metastatic germ cell tumour.
* Patients with a prior history of chemotherapy or radiotherapy at study entry.
* Prior history of thoracic surgery or significant chest trauma
* Prior history of significant smoking or respiratory disease.
* The presence of another malignancy, where the extent of disease or treatment for that condition may interfere with the study endpoints.
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule.
* Inability to lie flat for imaging.
* Contra-indications to receiving iodine-based contrast during thoracic CT - those with marked renal failure not on dialysis, known allergy to contrast medium, history of anaphylaxis, known or suspected thyroid carcinoma and inability to gain intra-venous access.
* Contraindications to MRI examination including indwelling pacemaker, non-MRI compatible metallic implant, severe claustrophobia, intra-ocular foreign body.
* Epilepsy requiring on-going medical treatment, or a seizure within the past year.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2012-04; Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Imaging parameters from MRI scan after inhalation of hyperpolarized xenon gas | Up to one year after first scan
  Maps of Apparent Diffusion Coefficient and objective measures of regional lung Production of Xe-129 ADC maps co-registered to CT and objective measures of regional lung anatomy, ventilation and perfusion in normals with hyperpolarized Xe-129 MR imaging (ADC quantification in cm2s-1). Derivation of reproducibility data

SECONDARY OUTCOMES:
To produce and confirm reliability of maps to show regional blood perfusion in the lung area | On entry to the study and one year later
  Maps of the dissolved fraction of Xe-129 to show hyperpolarized xenon transferred from the lungs to the blood
Repeatability of the 129-Xe MR scans | On study entry and one year later
  Compare scans on the same day with the patient prone and supine. Compare scans taken supine one year apart

CONTACTS AND LOCATIONS:
Overall Officials: Fergus V Gleeson, Principal Investigator — Oxford University Hospitals NHS Trust
Locations (1):
- Oxford University Hospitals NHS Trust, Oxford, England, United Kingdom